CLINICAL TRIAL: NCT04026022
Title: Perioperative Off-label Application (From Admission up to 72 Hours Postoperatively) of Fentanyl TTS as Part of a Pain Management in Comparison to a Certified Pain Medication Management in Adult Patients With a Hip Fracture.
Brief Title: Traumatologic Acute Pain Management With Fentanyl Transdermal Therapeutic System (TTS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2gas
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2019-07

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2)
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard pain management (Placebo Comparator): Besides the standard pain management a placebo TTS (normal wound plaster) will be administered in the Emergency Room (ER) or Post Anaesthesia Care Unit (PACU)
  Interventions: Drug: Placebo
- Modified pain management (Experimental): Patients will be treated perioperatively with a new pain management, that has been modified to integrate the 2017 ESA guidelines on prevention/treatment of postoperative delirium. Moreover patients will be administered a 12µg/h Fentanyl TTS in the ER or PACU. The ER TTS will only be administered if the patients still has mild to intense pain after initial i.v. treatment as well as reposition of the fractured hip. Further aspects of the modified management are: avoiding benzodiazepines, allowing oral fluids up to 2 hours before surgery, intraoperative monitoring of anaesthesia depth and at least 1,8 ltr crystalloid infusion per day
  Interventions: Drug: Fentanyl Transdermal System

INTERVENTIONS:
Drug: Fentanyl Transdermal System — Patients will be treated perioperatively with a new pain management, that has been modified to integrate the 2017 ESA guidelines on prevention/treatment of postoperative delirium. Moreover patients will be administered a 12µg/h Fentanyl TTS in the ER or PACU. The ER TTS will only be administered if the patients still has mild to intense pain after initial intravenous (i.v.) treatment as well as reposition of the fractured hip. Further aspects of the modified management are: avoiding benzodiazepines, allowing oral fluids up to 2 hours before surgery, intraoperative monitoring of anaesthesia depth and at least 1,8 ltr crystalloid infusion per day.
  Arms: Modified pain management
Drug: Placebo — Placebo plaster in the ER or PACU
  Arms: Standard pain management

SUMMARY:
Aim of the study is an examination whether a modified perioperative pain management system, that integrates the 2017 European Society of Anaesthesiology (ESA) guidelines for treatment of postoperative Delirium, can improve patient's wellbeing in comparison to the current certified standard management.

DETAILED DESCRIPTION:
Aim of the study is to evaluate whether the integration of the 2017 ESA guidelines for treatment of postoperative Delirium in a pain management, can improve patient's wellbeing in comparison to the current certified standard management. Adherence to the modified management includes minimizing nil per os time, renouncing benzodiazepines, 1.8 ltr crystalloid infusion per day, simplified standard medication option and postoperative 12µg/h Fentanyl TTS for 72h (for wound pain).

ELIGIBILITY:
Inclusion Criteria:

* adult patients with hip fractures that have to be operated (ICD S72.01-S72.2)

Exclusion Criteria:

* severe liver damage
* ongoing dialysis therapy
* Monoamine oxidase inhibitor intake
* inability to give consent to trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Patient's wellbeing in the awakening room | 1 year
  Wellbeing assessed with the "Anaesthesiological Questionnaire" (ANP) which is a self-rating method for the assessment of postoperative complaints and patient wellbeing. The rating scales from 0 to 3, with 0="none" and 3="strongly". Higher wellbeing values represent a better outcome.

SECONDARY OUTCOMES:
Complication rate (delirium, periprosthetic fractures, wound infections etc) | Through study completion, an average of 10 days
  All complications occuring during hospital stay will be statistically evaluated for differences between the two study groups.
Efficacy of the pain management in reducing pain | Through study completion, an average of 10 days
  Pain will be assessed with the (verbal) Numerical Rating Scale (NRS) and statistically evaluated for differences between the two study groups. NRS scales from 1 to 10, with 1 describing the lowest pain score and 10 the highest pain score. Lower NRS describes a better outcome.
Interview assessed identification of selfreported parameters influencing patient-wellbeing | Through study completion, an average of 72 hours postoperatively
  Feedback interviews with the patients giving them the opportunity to express what influenced their wellbeing the most.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Hospital LKH Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
After publication of our results, all collected data will be made available in respect of data privacy laws.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Labmayr V, Rief M, Reinbacher P, Gebauer D, Smigaj J, Sandner-Kiesling A, Papamargaritis V, Michaeli K, Bornemann-Cimenti H, Schittek GA. Simplified Pain Management Including Fentanyl TTS in PACU Patients With Hip Fracture Surgery to Improve Patients' Well-Being: A Double-Blind Randomized Trial. J Perianesth Nurs. 2024 Jun;39(3):461-467. doi: 10.1016/j.jopan.2023.10.004. Epub 2023 Dec 11. PMID 38085188